CLINICAL TRIAL: NCT02539394
Title: Do Intraoperative Topical Corticosteroids Aid in the Prevention of Postoperative Dysphagia Following Elective Anterior Cervical Discectomy and Fusion? A Randomized, Controlled, Double Blinded Clinical Trial
Brief Title: Effect of Topical Corticosteroids on Dysphagia in Anterior Cervical Discectomy and Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014-145
Record Dates: First submitted 2015-08-27; First posted 2015-09-03 (Estimated); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Cervical Disc Herniation; Cervical Degenerative Disc Disease; Cervical Spondylotic Myelopathy; Dysphagia; Osteoarthritis of Cervical Spine
Keywords: Anterior Cervical Discectomy and Fusion; Dysphagia; ACDF
MeSH Terms: conditions — Deglutition Disorders | interventions — Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Procedure: Anterior Cervical Discectomy and Fusion. The treatment arm will receive 40 mg of Methylprednisolone Acetate delivered with a Hemostatic Matrix Kit prior to closure.
  Interventions: Drug: Methylprednisolone Acetate; Other: Hemostatic Matrix Kit
- Control (Placebo Comparator): Procedure: Anterior Cervical Discectomy and Fusion. The control group will receive only a Hemostatic Matrix Kit prior to closure.
  Interventions: Other: Hemostatic Matrix Kit

INTERVENTIONS:
Drug: Methylprednisolone Acetate — Methylprednisolone Acetate is a corticosteroid known to reduce swelling and inflammation.
  Other Names: Depo-Medrol
  Arms: Treatment
Other: Hemostatic Matrix Kit — Hemostatic Matrix Kits help prevent uncontrollable bleeding in a operative site during a procedure.

SUMMARY:
The purpose of this study is to determine what effect intraoperative topical steroids have on reducing swallowing difficulty following Anterior Cervical Discectomy and Fusion surgery.

DETAILED DESCRIPTION:
Background: Dysphagia is a serious post-operative concern in patients following anterior cervical surgery. Although many experts have acknowledged that dysphagia is often incompletely understood and defined, there is a significant amount of literature to support the significance of this clinical entity. This is the first randomized study to examine the use of topical steroids for the prevention of dysphagia postoperatively after anterior cervical discectomy and fusion.

Study Design: This study is a single site, double blinded randomized control trial. All individuals undergoing 2-4 level ACDF that meet the inclusion criteria will be randomized to either:

1. treatment arm or
2. control arm.

Both arms will undergo their planned surgeries and will receive the exact same procedure and standard of care as if they were not enrolled in a study. The only difference is that the treatment arm will receive 40 mg of Methylprednisolone Acetate delivered with one Hemostatic Matrix Kit injectable delivery vehicle prior to closure in the prevertebral soft tissues. The control group will receive only Hemostatic Matrix Kit prior to closure in the prevertebral soft tissues.

Outcomes: Patients will be asked to fill out questionnaires that assess dysphagia, general swallowing difficulty, and how neck pain impacts their quality of life. Additionally Radiographic images will be obtained at set time points to evaluate soft tissue inflammation and bony fusion.

ELIGIBILITY:
Inclusion Criteria:

* Any patient > 18 years undergoing a 2-4 level Anterior Cervical Discectomy and Fusion

Exclusion Criteria:

* Patients undergoing revision surgery
* Pediatric patients
* Trauma patients with cervical spine fractures
* Patients with cancer
* Patients with active infection
* Patients with a known allergy to Methylprednisolone Acetate
* Patients who refuse to participate
* Non English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-08; Primary Completion 2020-11-12 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Albert, MD, Principal Investigator — Hospital for Special Surgery, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 64 | 64
Completed | 56 | 53
Not Completed | 8 | 11
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Incomplete dataset | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 56 | 53 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.5) | 58.4 (11.5) | 58.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 27 | 29 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 56 | 53 | 109
Smoking status [Count of Participants; unit: Participants]
  Not Applicable | 27 | 35 | 62
  Former (quit > 30 days) | 23 | 14 | 37
  Current (within the last 30 days) | 6 | 4 | 10
Diagnosis [Count of Participants; unit: Participants]
  Spondylosis | 39 | 32 | 71
  Herniated disc | 8 | 4 | 12
  Stenosis | 10 | 10 | 20
  Osteoarthritis of the Cervical Spine | 0 | 1 | 1
  Myelopathy | 14 | 14 | 28
  Radiculopathy | 31 | 23 | 54
  Myeloradiculopathy | 15 | 17 | 32
  Cervical disk disorder | 1 | 0 | 1
  Foraminal Stenosis | 1 | 6 | 7
  Disk degrative disease | 2 | 5 | 7
Charlson Comorbidities Index (CCI) [Median (Inter-Quartile Range); unit: index] — The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes found in administrative data, such as hospital abstracts data. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
  index | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Degree of Dysphagia Patients Experience (Burden)
Description: SWAL-QOL survey - Burden domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Analysis performed on patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 100 [100 to 100] | 100 [100 to 100]
  POD1 | 50 [25 to 87.5] | 75 [50 to 100]
  POD2 | 62.5 [25 to 87.5] | 75 [50 to 100]
  4-6 weeks | 100 [62.5 to 100] | 100 [100 to 100]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 100 [87.5 to 100] | 100 [100 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 100 [100 to 100] | 100 [100 to 100]
  1 year: number analyzed (Participants) | 47 | 48
  1 year | 100 [87.5 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Burden is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.394, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Burden is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.017, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD2 SWAL-QOL - Burden is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.015, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Burden is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.125, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Degree of Dysphagia Patients Experience (Eating Desire)
Description: SWAL-QOL survey - Eating desire domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 100 [100 to 100] | 100 [100 to 100]
  POD1 | 83.3 [58.3 to 100] | 87.5 [60.4 to 100]
  POD2 | 83.3 [58.3 to 100] | 91.7 [68.75 to 100]
  4-6 weeks | 100 [83.3 to 100] | 100 [100 to 100]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 100 [100 to 100] | 100 [100 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 100 [100 to 100] | 100 [100 to 100]
  1 year: number analyzed (Participants) | 47 | 48
  1 year | 100 [100 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Eating desire is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.043, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Eating desire is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.606, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD2 SWAL-QOL - Eating desire is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.155, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Eating desire is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.019, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Degree of Dysphagia Patients Experience (Eating Duration)
Description: SWAL-QOL survey - Eating duration domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 100 [100 to 100] | 100 [100 to 100]
  POD1 | 75 [25 to 93.75] | 75 [37.5 to 100]
  POD2 | 50 [18.75 to 87.5] | 75 [37.5 to 100]
  4-6 weeks | 87.5 [43.75 to 100] | 100 [75 to 100]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 100 [75 to 100] | 100 [87.5 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 100 [87.5 to 100] | 100 [100 to 100]
  1 year: number analyzed (Participants) | 47 | 48
  1 year | 100 [87.5 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Eating duration is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.250, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Eating duration is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.478, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control; The distribution of POD2 SWAL-QOL - Eating duration is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.019, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Eating duration is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.049, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Degree of Dysphagia Patients Experience (Food Selection)
Description: SWAL-QOL survey - Food Selection domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 100 [100 to 100] | 100 [100 to 100]
  POD1 | 75 [37.5 to 93.75] | 93.75 [50 to 100]
  POD2 | 62.5 [25 to 100] | 75 [62.5 to 100]
  4-6 weeks | 100 [75 to 100] | 100 [75 to 100]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 100 [100 to 100] | 100 [100 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 100 [100 to 100] | 100 [100 to 100]
  1 year: number analyzed (Participants) | 47 | 47
  1 year | 100 [100 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Food selection is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.376, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Food selection is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.013, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD2 SWAL-QOL - Food selection is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.049, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Food selection is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.300, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Degree of Dysphagia Patients Experience (Communication)
Description: SWAL-QOL survey - Communication domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 100 [100 to 100] | 100 [100 to 100]
  POD1 | 100 [81.25 to 100] | 100 [87.5 to 100]
  POD2 | 100 [75 to 100] | 100 [90.625 to 100]
  4-6 weeks | 100 [75 to 100] | 100 [100 to 100]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 100 [100 to 100] | 100 [100 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 100 [100 to 100] | 100 [100 to 100]
  1 year: number analyzed (Participants) | 47 | 48
  1 year | 100 [100 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Communication is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.037, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Communication is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.858, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD2 SWAL-QOL - Communication is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.042, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Communication is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.031, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Degree of Dysphagia Patients Experience (Fear Swallow)
Description: SWAL-QOL survey - Fear swallow domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 100 [100 to 100] | 100 [100 to 100]
  POD1 | 93.75 [75 to 100] | 100 [87.5 to 100]
  POD2 | 87.5 [56.25 to 100] | 100 [76.6 to 100]
  4-6 weeks | 93.75 [84.4 to 100] | 100 [87.5 to 100]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 100 [87.5 to 100] | 100 [100 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 100 [93.75 to 100] | 100 [100 to 100]
  1 year: number analyzed (Participants) | 47 | 48
  1 year | 100 [87.5 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Fear swallow is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.343, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Fear swallow is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.022, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD2 SWAL-QOL - Fear swallow is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.018, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Fear swallow is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.008, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Degree of Dysphagia Patients Experience (Social)
Description: SWAL-QOL survey - Social domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 100 [100 to 100] | 100 [100 to 100]
  POD1 | 95 [67.5 to 100] | 100 [75 to 100]
  POD2 | 85 [25 to 100] | 100 [56.25 to 100]
  4-6 weeks | 100 [85 to 100] | 100 [95 to 100]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 100 [100 to 100] | 100 [100 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 100 [100 to 100] | 100 [100 to 100]
  1 year: number analyzed (Participants) | 47 | 48
  1 year | 100 [100 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Social is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.280, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Social is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.483, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD2 SWAL-QOL - Social is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.070, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Social is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.200, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Degree of Dysphagia Patients Experience (Mental)
Description: SWAL-QOL survey - Mental domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 100 [100 to 100] | 100 [100 to 100]
  POD1 | 80 [50 to 100] | 100 [75 to 100]
  POD2 | 85 [50 to 100] | 97.5 [70 to 100]
  4-6 weeks | 95 [77.5 to 100] | 100 [80 to 100]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 100 [85 to 100] | 100 [100 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 100 [95 to 100] | 100 [100 to 100]
  1 year: number analyzed (Participants) | 47 | 48
  1 year | 100 [90 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Mental is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.148, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Mental is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.040, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD2 SWAL-QOL - Mental is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.042, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Mental is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.319, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Degree of Dysphagia Patients Experience (Sleep)
Description: SWAL-QOL survey - Sleep domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 75 [50 to 100] | 81.25 [62.5 to 100]
  POD1 | 62.5 [37.5 to 75] | 56.25 [37.5 to 87.5]
  POD2 | 50 [25 to 75] | 62.5 [50 to 75]
  4-6 weeks | 50 [37.5 to 81.25] | 75 [50 to 87.5]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 62.5 [50 to 87.5] | 75 [62.5 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 62.5 [50 to 100] | 75 [62.5 to 100]
  1 year: number analyzed (Participants) | 47 | 48
  1 year | 75 [50 to 87.5] | 87.5 [50 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Sleep is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.161, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Sleep is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.763, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD2 SWAL-QOL - Sleep is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.178, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Sleep is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.091, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Degree of Dysphagia Patients Experience (Fatigue)
Description: SWAL-QOL survey - Fatigue domain Score ranges between 0 and 100 (worst-best)
Time Frame: Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative | 83.33 [54.17 to 100] | 83.33 [60.42 to 100]
  POD1 | 58.33 [25 to 70.83] | 58.33 [25 to 83.33]
  POD2 | 58.33 [33.33 to 75] | 66.67 [41.67 to 83.33]
  4-6 weeks | 58.33 [41.67 to 75] | 75 [58.33 to 97.92]
  3 months: number analyzed (Participants) | 51 | 53
  3 months | 75 [58.33 to 91.67] | 83.33 [70.83 to 100]
  6 months: number analyzed (Participants) | 51 | 51
  6 months | 75 [58.33 to 91.67] | 83.33 [66.67 to 100]
  1 year: number analyzed (Participants) | 47 | 48
  1 year | 75 [66.67 to 91.67] | 91.67 [66.67 to 100]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative SWAL-QOL - Fatigue is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.602, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of POD1 SWAL-QOL - Fatigue is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.302, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD2 SWAL-QOL - Fatigue is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.114, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of 4-6 weeks SWAL-QOL - Fatigue is the same across the 2 arms; Test type: Equivalence — 43 patient in each group need to achieved >80% power to detect a 15 point differences in SWAL-QOL survey; p = 0.005, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Patient Reported Swallowing Difficulty Over 1 Year
Description: The Eating Assessment Tool (EAT-10) is used to screen for self-perceived oropharyngeal dysphagia (OD) in community-dwelling elders. A summated EAT-10 total score ranges from 0 to 40, with a score ≥ 3 indicative of OD.
  Modified Eat-10 : Eat-10 questionnaire without questions 1 ("My swallowing problem has caused me to lose weight") and 2 ("My swallowing problem interferes with my ability to go out for meals") to be applicable during hospitalization.
  Eat-10 interpretation: Score ranging from 0 to 40 (best-worst)
  * each question response is 0-4, 0=no problem and 4=severe problem; score is a summation of each question's response Modified EAT-10 interpretation: Score ranging from 0 to 32 (best-worst)
  * each question response is 0-4, 0=no problem and 4=severe problem; score is a summation of each question's response
Time Frame: Pre-Op, Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
score on a scale
  Pre-operative Eat-10 | 0 [0 to 0] | 0 [0 to 0]
  Pre-operative Eat-10 modified | 0 [0 to 0] | 0 [0 to 0]
  POD1 Eat-10 | 16 [7 to 19.5] | 9 [4.25 to 20.75]
  POD1 Eat-10 modified | 14 [7 to 19.5] | 8.5 [4 to 18]
  POD2 Eat-10 | 16 [7 to 25.5] | 8 [3.25 to 21.75]
  POD2 Eat-10 modified | 14 [7 to 20.5] | 7 [3 to 17.75]
  4-6 weeks Eat-10 | 5 [0 to 11.5] | 2 [0 to 6]
  4-6 weeks Eat-10 modified | 4 [0 to 9.5] | 2 [0 to 5]
  3 months Eat-10: number analyzed (Participants) | 51 | 53
  3 months Eat-10 | 2 [0 to 6] | 0 [0 to 4]
  3 months Eat-10 modified: number analyzed (Participants) | 51 | 53
  3 months Eat-10 modified | 2 [0 to 6] | 0 [0 to 4]
  6 months Eat-10: number analyzed (Participants) | 51 | 51
  6 months Eat-10 | 1 [0 to 5] | 0 [0 to 2]
  6 months Eat-10 modified: number analyzed (Participants) | 51 | 51
  6 months Eat-10 modified | 1 [0 to 4] | 0 [0 to 2]
  1 year Eat-10: number analyzed (Participants) | 47 | 48
  1 year Eat-10 | 0 [0 to 5] | 0 [0 to 2]
  1 year Eat-10 modified: number analyzed (Participants) | 47 | 48
  1 year Eat-10 modified | 0 [0 to 5] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Control vs Treatment; The distribution of Pre-operative Eat-10 is the same across the 2 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.933, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Treatment; The distribution of Pre-operative modified Eat-10 is the same across the 2 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.950, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Treatment; The distribution of POD1 Eat-10 is the same across the 2 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.059, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Treatment; The distribution of POD1 modified Eat-10 is the same across the 2 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.042, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Control vs Treatment; The distribution of POD2 Eat-10 is the same across the 2 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.032, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Control vs Treatment; The distribution of POD2 modified Eat-10 is the same across the 2 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.014, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Control vs Treatment; The distribution of 4-6 weeks Eat-10 is the same across the 2 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.030, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Control vs Treatment; The distribution of 4-6 weeks modified Eat-10 is the same across the 2 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.039, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Patients' Bazaz Dysphagia Score - Liquid
Description: Bazaz dysphagia scale defines dysphagia as none, mild, moderate and severe, depending on patients' symptoms with solid and liquid foods.
Time Frame: Pre-Op, Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
Participants
  Pre-operative: None | 47 | 54
  Pre-operative: Rare | 6 | 2
  POD1: None | 20 | 36
  POD1: Rare | 33 | 20
  POD2: number analyzed (Participants) | 51 | 54
  POD2: None | 17 | 23
  POD2: Rare | 34 | 31
  6-4 weeks: None | 35 | 39
  6-4 weeks: Rare | 18 | 17
  3 months: number analyzed (Participants) | 50 | 52
  3 months: None | 39 | 39
  3 months: Rare | 11 | 13
  6 months: number analyzed (Participants) | 51 | 51
  6 months: None | 42 | 41
  6 months: Rare | 9 | 10
  1 year: number analyzed (Participants) | 45 | 47
  1 year: None | 35 | 40
  1 year: Rare | 10 | 7
Statistical Analysis 1: Comparison: Control; Proportion of Pre-operative Bazaz Liquid is the same between the 2 arms; Test type: Equivalence — Two-sided; p = 0.121, Chi-squared
Statistical Analysis 2: Comparison: Control vs Treatment; Proportion of POD1 Bazaz Liquid is the same between the 2 arms; Test type: Equivalence — Two-sided; p = 0.006, Chi-squared
Statistical Analysis 3: Comparison: Control vs Treatment; Proportion of POD2 Bazaz Liquid is the same between the 2 arms; Test type: Equivalence — Two-sided; p = 0.329, Chi-squared
Statistical Analysis 4: Comparison: Control vs Treatment; Proportion of 4-6 weeks Bazaz Liquid is the same between the 2 arms; Test type: Equivalence — Two-sided; p = 0.687, Chi-squared

13. Secondary Outcome: Patients' Bazaz Dysphagia Score - Solid
Description: as for outcome 12
Time Frame: Pre-Op, Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
Participants
  Pre-operative: None | 44 | 52
  Pre-operative: Rare | 8 | 2
  Pre-operative: Occasionally (only with specific food) | 0 | 2
  Pre-operative: Frequent (majority of solids) | 1 | 0
  POD1: None | 9 | 17
  POD1: Rare | 8 | 11
  POD1: Occasionally (only with specific food) | 21 | 18
  POD1: Frequent (majority of solids) | 15 | 10
  POD2: number analyzed (Participants) | 51 | 54
  POD2: None | 6 | 15
  POD2: Rare | 9 | 13
  POD2: Occasionally (only with specific food) | 19 | 15
  POD2: Frequent (majority of solids) | 17 | 11
  6-4 weeks: None | 18 | 27
  6-4 weeks: Rare | 18 | 16
  6-4 weeks: Occasionally (only with specific food) | 11 | 11
  6-4 weeks: Frequent (majority of solids) | 6 | 2
  3 months: number analyzed (Participants) | 50 | 52
  3 months: None | 25 | 34
  3 months: Rare | 11 | 8
  3 months: Occasionally (only with specific food) | 12 | 10
  3 months: Frequent (majority of solids) | 2 | 0
  6 months: number analyzed (Participants) | 51 | 51
  6 months: None | 30 | 37
  6 months: Rare | 15 | 10
  6 months: Occasionally (only with specific food) | 5 | 3
  6 months: Frequent (majority of solids) | 1 | 1
  1 year: number analyzed (Participants) | 45 | 47
  1 year: None | 29 | 35
  1 year: Rare | 7 | 6
  1 year: Occasionally (only with specific food) | 9 | 4
  1 year: Frequent (majority of solids) | 0 | 2
Statistical Analysis 1: Comparison: Control vs Treatment; Proportion of Pre-operative Bazaz Solid is the same between the 2 arms; Test type: Equivalence — Two-sided; p = 0.066, Chi-squared
Statistical Analysis 2: Comparison: Control vs Treatment; Proportion of POD1 Bazaz Solid is the same between the 2 arms; Test type: Equivalence — Two-sided; p = 0.252, Chi-squared
Statistical Analysis 3: Comparison: Control vs Treatment; Proportion of POD2 Bazaz Solid is the same between the 2 arms; Test type: Equivalence — Two-sided; p = 0.100, Chi-squared
Statistical Analysis 4: Comparison: Control vs Treatment; Proportion of 4-6 weeks Bazaz Solid is the same between the 2 arms; Test type: Equivalence — Two-sided; p = 0.279, Chi-squared

14. Secondary Outcome: Patients' Neck Disability
Description: Neck Disability Index (NDI) Range from 0 to 100 (best-worst)
Time Frame: Pre-Op, Week 4-6, 3 Months, 6 Months, 12 Months
Population: People with completed follow-up
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
index
  Pre-operative: number analyzed (Participants) | 51 | 55
  Pre-operative | 35.5 (20.1) | 29.9 (19.4)
  4-6 weeks: number analyzed (Participants) | 51 | 54
  4-6 weeks | 35.3 (17.5) | 30.8 (20.6)
  3 months: number analyzed (Participants) | 50 | 50
  3 months | 27.3 (15.8) | 17.7 (14.3)
  6 months: number analyzed (Participants) | 51 | 50
  6 months | 23.9 (17.7) | 15.4 (13.8)
  1 year: number analyzed (Participants) | 47 | 46
  1 year | 20.6 (17.9) | 13.2 (12.0)
Statistical Analysis 1: Comparison: Control vs Treatment; The means Pre-operative NDI for the two populations is equal; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.145, t-test, 2 sided
Statistical Analysis 2: Comparison: Control vs Treatment; The means 4-6 weeks NDI for the two populations is equal; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.234, t-test, 2 sided

15. Secondary Outcome: Patients' Pain Scores on the Visual Analog Scale - Neck Pain
Description: Visual Analog Scale (VAS) - Neck pain Range from 0 to 100 (best-worst)
Time Frame: Pre-Op, Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
units on a scale
  Pre-operative: number analyzed (Participants) | 51 | 55
  Pre-operative | 54.5 [22.5 to 70] | 26 [5.8 to 61.5]
  POD1: number analyzed (Participants) | 47 | 54
  POD1 | 51.5 [25 to 77] | 48.25 [8.025 to 61.125]
  POD2: number analyzed (Participants) | 47 | 52
  POD2 | 51 [21.5 to 69] | 26.5 [11.5 to 49.125]
  4-6 weeks: number analyzed (Participants) | 51 | 53
  4-6 weeks | 20 [5.5 to 40] | 14.5 [4.5 to 30.25]
  3 months: number analyzed (Participants) | 51 | 51
  3 months | 22 [5 to 49] | 9.5 [2 to 25]
  6 months: number analyzed (Participants) | 51 | 48
  6 months | 14 [5.5 to 45] | 6 [1.5 to 19.375]
  1 year: number analyzed (Participants) | 46 | 48
  1 year | 12.25 [0.7 to 52.125] | 6.5 [0.875 to 14.125]

16. Secondary Outcome: Patients' Pain Scores on the Visual Analog Scale - Left Arm Pain
Description: Visual Analog Scale (VAS) - Left arm pain Range from 0 to 100 (best-worst)
Time Frame: Pre-Op, Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
units on a scale
  Pre-operative | 17.5 [1 to 52] | 19 [2.1 to 53.9]
  POD1 | 10 [0 to 38] | 5.35 [0 to 17]
  POD2 | 5 [0 to 38] | 6.45 [0 to 16.5]
  4-6 weeks | 6.45 [0 to 28] | 2.75 [0.125 to 13]
  3 months | 5.8 [0 to 16] | 2.5 [0 to 16]
  6 months | 2 [0 to 17.5] | 1.175 [0 to 11]
  1 year | 4 [0 to 21.5] | 1 [0 to 8]

17. Secondary Outcome: Patients' Pain Scores on the Visual Analog Scale - Right Arm Pain
Description: Visual Analog Scale (VAS) - Right arm pain Range from 0 to 100 (best-worst)
Time Frame: Pre-Op, Post-Op Day 1, Post-Op Day 2, Week 4-6, 3 Months, 6 Months, 12 Months
Population: Patient with completed follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
units on a scale
  Pre-operative: number analyzed (Participants) | 51 | 55
  Pre-operative | 20 [2 to 67] | 15.5 [0 to 38.4]
  POD1: number analyzed (Participants) | 47 | 54
  POD1 | 2 [0 to 20.5] | 2.25 [0 to 10]
  POD2: number analyzed (Participants) | 47 | 52
  POD2 | 3 [0 to 22] | 4 [0 to 16]
  4-6 weeks: number analyzed (Participants) | 51 | 53
  4-6 weeks | 7 [0 to 32] | 2 [0 to 11.9]
  3 months: number analyzed (Participants) | 51 | 51
  3 months | 4 [0 to 30] | 2 [0 to 15]
  6 months: number analyzed (Participants) | 51 | 48
  6 months | 6 [0 to 40] | 2 [0 to 8]
  1 year: number analyzed (Participants) | 46 | 47
  1 year | 3.5 [0 to 26.25] | 2.4 [0 to 9]

18. Secondary Outcome: Change in Pre-vertebral Soft Tissue Swelling Over 1 Year
Description: We are unable to report this outcome measure because soft tissue swelling was not assessed. The PI deemed it would not be included for this study as there is not a clinical or research standard to do so, nor is there normative data over time to compare against. Thus, data were not collected.
Time Frame: Pre-Op, Post-Op Day 1, Week 4-6, 3 Months, 6 Months, 12 Months
Population: We are unable to report this outcome measure because soft tissue swelling was not assessed. The PI deemed it would not be included for this study as there is not a clinical or research standard to do so, nor is there normative data over time to compare against.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Fusion Rate
Description: 1. Flex-Ex X-rays
  2. Bony bridging on a CT scan
  3. Obvious bony remodeling on lateral X-ray
Time Frame: 12 Months
Population: Subjects with 12 month follow up visit with X-rays. All others were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 50 | 45
Participants | 25 | 23
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.99, Fisher Exact

20. Secondary Outcome: Adverse Event
Description: Adverse Event (AE) following surgical treatment.
  Adverse event were classified by severity based on the AO-ISSG criteria and treatment required:
  Mild: Observed, medication, consult, X-ray. Essentially any management that was quick and easy and could be done at bedside Moderate: ICU admission, re-intubation, complication that had a documented prolonged hospital stay, medical procedure (such as flexible endoscopy), re-presentation to ED Severe: Inpatient re-admission, return to OR for any reason, mortality, failed OR.
  AE were also categorize as Surgery-site related or unrelated adverse event. Finally, AE were also categorize as potentially related to steroid use (example: leukocytosis, pseudoarthrosis, or wound complications)
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 53 | 56
Participants
  Any Adverse Event? | 44 | 47
  Mild/Moderate Adverse Event? | 42 | 46
  Severe Adverse Event? | 3 | 3
  Adverse Event Related to Operated Site? | 38 | 38
  Adverse Event Unrelated to Operated Site? | 26 | 30
  Mild/Moderate Adverse Event Related to Operated Site? | 36 | 37
  Mild/Moderate Adverse Event Unrelated to Operated Site? | 26 | 30
  Severe Adverse Event Related to Operated Site? | 3 | 3
  Severe Adverse Event Unrelated to Operated Site? | 0 | 0
  Adverse Event Potentially Related to Steroid Use? | 11 | 16
  Adverse Event Unrelated to Steroid use? | 43 | 42
  Mild/Moderate Adverse Event Potentially Related to Steroid Use? | 9 | 15
  Mild/Moderate Adverse Event Unrelated to Steroid use? | 42 | 41
  Severe Adverse Event Potentially Related to Steroid Use? | 2 | 1
  Severe Adverse Event Unrelated to Steroid use? | 1 | 2

ADVERSE EVENTS:
Time Frame: 12 months
Description: For standardization for mild-mod-severe AE was mostly based on the AO-ISSG criteria:
  Mild: Observed, medication, consult, X-ray. Essentially any management that was quick and easy and could be done at bedside Moderate: ICU admission, re-intubation, complication that had a documented prolonged hospital stay, medical procedure (such as flexible endoscopy), re-presentation to ED Severe: Inpatient re-admission, return to OR for any reason, mortality, failed OR.
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/56
Serious Adverse Events (participants affected / at risk) | 3/53 | 3/56
Other Adverse Events (participants affected / at risk) | 42/53 | 46/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=53) | Treatment (N=56)
GastroIntestinal (Gastrointestinal disorders) | 0 | 1 — Constipation, Dysphagia, Nausea / Vomiting, Reflux
Skeletal (Musculoskeletal and connective tissue disorders) | 3 | 2 — Hardware Complication, Pseudoarthrosis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=53) | Treatment (N=56)
Cardiovascular (Cardiac disorders) | 17 | 15 — ABLA, Acute Cardiac, Arrhythmia, DVT, Hyperkalemia, Hypertension, Hyponatremia, Hypotension/Hypovolemia, Leukocytosis, VTE
Digestive (General disorders) | 1 | 0 — Dysphagia
Endocrine (Endocrine disorders) | 0 | 6 — Hyperglycemia
Genitourinary (Reproductive system and breast disorders) | 1 | 0 — Urinary Retention
Gastrointestinal (Gastrointestinal disorders) | 24 | 23 — Constipation, Dysphagia, Nausea / Vomiting, Reflux
Hematologic (Blood and lymphatic system disorders) | 7 | 9 — Leukocytosis
Immune (Immune system disorders) | 1 | 1
Integumentary (Skin and subcutaneous tissue disorders) | 2 | 1
Neurologic (Nervous system disorders) | 1 | 3 — Dizziness/Vertigo, Migraine
Pain (General disorders) | 19 | 28 — Non-Radicular, Radicular
Respiratory (Respiratory, thoracic and mediastinal disorders) | 10 | 6 — Aspiration, Atelectasis, Hypoxia
Skeletal (Musculoskeletal and connective tissue disorders) | 0 | 0 — Hardware Complication, Pseudoarthrosis
Wound (Surgical and medical procedures) | 5 | 3 — Hematoma, Infection, SSI

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT02539394/Prot_SAP_000.pdf
  • Informed Consent Form (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT02539394/ICF_001.pdf